CLINICAL TRIAL: NCT06139354
Title: Pilot Testing of a Patient-provider Decision Aid for HIV Post-exposure Prophylaxis Following Sexual Assault
Brief Title: Patient-provider Decision Aid for HIV Post-exposure Prophylaxis Following Sexual Assault
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: University of California, Davis (Other); District of Columbia Forensic Nurse Examiners (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 276376
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Hiv
Keywords: sexual assault
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- decision aid (Experimental): A digital, interactive patient-provider HIV PEP decision aid. The decision aid will incorporate five sections of content: 1) key clinical factors input by providers; 2) tailored HIV risk sharing information; 3) standardized multimedia educational messaging regarding the effectiveness, risks, and benefits of HIV PEP; 4) direct comparisons of priorities (e.g., physical well-being - "I want to do everything I can to prevent HIV," privacy - "I don't want others to know about the exposure," or cost - "I can't afford the pills'') completed by patients; and 5) tailored feedback regarding patient priorities for use in shared clinical decision making.
  Interventions: Behavioral: decision aid

INTERVENTIONS:
Behavioral: decision aid — A digital, interactive patient-provider HIV PEP decision aid. The decision aid will incorporate five sections of content: 1) key clinical factors input by providers; 2) tailored HIV risk sharing information; 3) standardized multimedia educational messaging regarding the effectiveness, risks, and benefits of HIV PEP; 4) direct comparisons of priorities (e.g., physical well-being - "I want to do everything I can to prevent HIV," privacy - "I don't want others to know about the exposure," or cost - "I can't afford the pills'') completed by patients; and 5) tailored feedback regarding patient priorities for use in shared clinical decision making.

SUMMARY:
The goal of this trial is to pilot a digital, interactive patient-provider HIV PEP decision aid. The decision aid will incorporate five sections of content: 1) key clinical factors input by providers; 2) tailored multimedia-based HIV risk sharing information; 3) standardized multimedia educational messaging regarding the effectiveness, risks, and benefits of HIV PEP; 4) direct comparisons of priorities (e.g., physical well-being - "I want to do everything I can to prevent HIV," privacy - "I don't want others to know about the exposure," or cost - "I can't afford the pills'') completed by patients; and 5) tailored feedback regarding patient priorities for use in shared clinical decision making.

DETAILED DESCRIPTION:
HIV post-exposure prophylaxis (PEP) decision-making following nonoccupational exposures (e.g. sexual assault, intravenous drug use (IVDU), consensual condomless sex) is a complicated clinical dilemma for patients and providers. HIV PEP is a highly effective course of antiretroviral medications taken for 28 days after an exposure. The estimated cost of lifetime HIV treatment is $326,000,3 and HIV PEP is cost effective for high risk exposures. Each year approximately 300,000 people in the US are sexually assaulted. For those who present for acute medical care following sexual assault, discussing HIV PEP is recommended by the International Association of Forensic Nurses (IAFN), Association of Nurses in AIDS Care, World Health Organization (WHO), and Department of Justice (DOJ).8-10 Despite its efficacy and these recommendations, HIV PEP remains inconsistently offered and initiated in sexual assault patient population.

Patient's must decide to take HIV PEP within 72 hours of an exposure. HIV PEP is not effective when initiated more than 72 hours after a potential exposure. These are not ideal conditions for making complex decisions. Patients report discussions regarding potential HIV exposure following sexual assault can cause an emotional response and asked providers to "do more" regarding explaining the realities of daily HIV PEP. Patients in the investigators' prior and ongoing work described inconsistent provider communication on the need for HIV PEP and lack of clarity regarding HIV risk as main barriers to decision making.

Provider HIV PEP provision patterns indicate important inequities in post-sexual assault HIV PEP patient care. The Centers for Disease Control and Prevention (CDC) guidelines include recommendations for HIV PEP following a non-occupational exposure, however there is a large gray area: decisions should be made on a "case-by-case" basis when the HIV status of the source is unknown. This translates into variations in clinical practice. Studies examining providers' behavior in offering HIV PEP to patients following sexual assault indicate they are influenced by factors such as pre-existing relationship between patient and the perpetrator, patient age, patient and perpetrator race, and anticipated patient financial burden. Additionally, in a survey previously conducted by the investigators, Sexual Assault Nurse Examiner (SANE) program coordinators reported a perception that patients "don't, won't, or can't follow-up" as a key reason for not offering HIV PEP routinely.

While not examined in HIV PEP, decision aids facilitate patient-provider communication and decision making. A 2017 Cochrane review of decision aids found patients who used a decision aid felt more informed about their decision and reported less decisional conflict. Patient-provider communication also improved.

Therefore, the goal of this pilot test a digital, interactive patient-provider HIV PEP decision aid. The decision aid will incorporate five sections of content: 1) key clinical factors input by providers; 2) tailored multimedia-based HIV risk sharing information; 3) standardized multimedia educational messaging regarding the effectiveness, risks, and benefits of HIV PEP; 4) direct comparisons of priorities (e.g., physical well-being - "I want to do everything I can to prevent HIV," privacy - "I don't want others to know about the exposure," or cost - "I can't afford the pills'') completed by patients; and 5) tailored feedback regarding patient priorities for use in shared clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* seeking care from DCFNE following sexual assault
* able to provide consent and participate in the study in English
* meets CDC criteria for HIV PEP [a) seeking care within 72 hours of potential exposure, b) potential exposure]

Exclusion Criteria:

* <18 years old
* Does not meet CDC criteria for HIV PEP [seeking care >72 hours after assault, assault with minimal/low exposure risk]
* unable to complete study requirements in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
decisional conflict | immediately post-intervention
  Modified questions from the Decisional Conflict Scale (O'Connor, 1993; 2010) as a measure of decision process. This scale tests whether using the HIV PEP decision aid helps a patient understand their options. This measure has a test-retest reliability from 0.75 to 0.81 and internal consistency (α) ranging from 0.72 to 0.92. The psychometric properties have been evaluated for the low literacy English version.
  Scores range from 0 [no decisional conflict] to 100 [very high decisional conflict].
decisional conflict | one month follow up
  Modified questions from the Decisional Conflict Scale (O'Connor, 1993; 2010) as a measure of decision process. This scale tests whether using the HIV PEP decision aid helps a patient understand their options. This measure has a test-retest reliability from 0.75 to 0.81 and internal consistency (α) ranging from 0.72 to 0.92. The psychometric properties have been evaluated for the low literacy English version.
  Scores range from 0 [no decisional conflict] to 100 [very high decisional conflict].

SECONDARY OUTCOMES:
HIV PEP acceptance | immediately post-intervention
  yes or no - patient decision to take or not take HIV PEP
HIV PEP completion | one month follow up
  Number of days (0-28) of HIV PEP patient completed
HIV PEP knowledge | immediately post-intervention
  Summary score from 6 items such as: "Within how long after an HIV exposure should PEP be started to prevent HIV?" & "How long do you take PEP?". Scores range from 0 to 6 based on the number of correct answers. Higher scores indicate more knowledge of HIV PEP. Items from Koblin et al. 2018.
HIV PEP knowledge | one month follow up
  Summary score from 6 items such as: "Within how long after an HIV exposure should PEP be started to prevent HIV?" & "How long do you take PEP?". Scores range from 0 to 6 based on the number of correct answers. Higher scores indicate more knowledge of HIV PEP. Items from Koblin et al. 2018.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Anderson, Principal Investigator — UAMS
Locations (1):
- District of Columbia Forensic Nurse Examiners, Washington D.C., District of Columbia, United States